CLINICAL TRIAL: NCT06734013
Title: Transcriptomics as an Aid in the Histological Diagnosis of Acute Rejection After Liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OLTpanel_2024; 2023.0189 (Other Grant/Funding Number: Fondazione Cassa di Risparmio in Bologna)
Record Dates: First submitted 2024-12-01; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Rejection; Transplant, Liver
Keywords: Liver transplant
MeSH Terms: conditions — Rejection, Psychology | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with post-OLT rejection (Experimental): The patient will be enrolled in a single visit, as per standard of care, clinical and general data will be collected and the biopsy will be performed
  Interventions: Diagnostic Test: Molecular diagnostic

INTERVENTIONS:
Diagnostic Test: Molecular diagnostic — RNA will be analysed using a Real-Time PCR expression card (TaqMan Real-Time PCR assay technology - Thermo Fisher Scientific). The analysis will be performed using a Real-Time Light Cycler 480 (Roche). The expression card will be customised for the study, including the genes cxcl9/10, cav-1, rhoj, cdh5, cd96, tnfsf8, il-21r, vcam, klrk1

SUMMARY:
The primary objective of this exploratory study is to identify genes associated with acute rejection in liver transplant patients. To this end, a panel of acute rejection indicator genes (both humoral and cell-mediated) will be selected from results published in the literature and applied to biological material derived from biopsies. The secodnary objective is to identify genes associated with the diagnosis of humoral acute rejection and those associated with the diagnosis of cell-mediated acute rejection.

DETAILED DESCRIPTION:
The possibility of introducing molecular diagnostics in support of histological and clinical diagnostics (still not routinely applied today but recommended by the most recent guidelines) will result in faster and more precise diagnostics, capable of highlighting early activation of cellular signals related to rejection in the absence yet of a frank clinical and histological picture. This will lead to a better diagnostic stratification of these patients, with the possibility of rationalising the choice of therapy.

AIMS: The primary objective of this exploratory study is to identify genes associated with acute rejection in liver transplant patients. To this end, a panel of acute rejection indicator genes (both humoral and cell-mediated) will be selected from published results in the literature and applied to biological material derived from biopsies. The secodnary objective is to identify genes associated with the diagnosis of humoral acute rejection and those associated with the diagnosis of cell-mediated acute rejection.

ENDPOINT/S: diagnostic (No of cases) of acute rejection; possible specific diagnosis of acute cell-mediated and humoral rejection.

STUDY DESIGN: The study is single-centre, observational, tissue-based, cross-sectional, exploratory, retrospective and prospective. Approximately 40 patients are expected to be enrolled, 20 retrospective and 20 prospective. All patients will be treated according to clinical practice: clinical and histological data will be collected in pseudonymous form. Routine histological and immunohistochemical investigations as well as RT-PCR analysis will be performed on the biopsy tissue (FFPE material). To assess the diagnostic sensitivity with regard to rejection status, and for panel development, a retrospective cohort of consecutive cases with acute rejection will be enrolled; for the prospective cohort, consecutive patients requiring liver biopsy for diagnostic indications will be enrolled.

STUDY POPULATION: The study will enrol patients undergoing OLT who require a liver biopsy for diagnostic indications. There is no restriction of sex or underlying pathology. Retrospective case enrolment is planned within the first 6 months of 2024. Prospective case enrolment will take place during 2024. Patients will be enrolled at the U.O. of Internal Medicine for the Treatment of Severe Organ Failures, IRCCS - Azienda Ospedaliero-Universitaria di Bologna Policlinico di S. Orsola, where the biopsy will be performed as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of post-OLT rejection prior to the visit at which they will be enrolled, with tissue available for RT-PCR investigations
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Identification of genes associated with acute rejection liver transplant. | At the time of biopsy, up to 6 months
  A panel of acute rejection indicator genes (both humoral and cell-mediated) will be selected from Scientific literature and applied to biological material from biopsies

SECONDARY OUTCOMES:
Identification of genes associated with the diagnosis of acute humoral rejection | At the time of biopsy, up to 6 months
  A panel of acute rejection indicator genes applied to biological material from biopsies
Identification of genes associated with the diagnosis of acute cell-mediated rejection | At the time of biopsy, up to 6 months
  A panel of acute rejection indicator genes applied to biological material from biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Malvi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No